CLINICAL TRIAL: NCT04921514
Title: Psychological Sequelae After Sudden Cardiac Death in the Patient and His Relatives
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/44
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder; Resuscitated Sudden Cardiac Death
Keywords: Sudden cardiac death
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: 40 participants (20 patients and 20 relatives)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient and relatives (Experimental)
  Interventions: Behavioral: SASRQ questionnaire; Behavioral: PCL-5 with LEC-5 questionnaire

INTERVENTIONS:
Behavioral: SASRQ questionnaire — During an interview with a trained psychologist, the presence of acute stress will be assessed by the SASRQ test within one week of the occurrence of a sudden recovered death.
  The diagnosis of acute post-traumatic stress disorder is made according to the presence of at least three dissociative symptoms out of five, and other symptoms of re-experiencing, avoidance or marked anxiety or hypervigilance. Each symptom is thus evaluated dichotomously. A symptom is present if the intensity of the response is 3 or more (0 "from 0 to 2" and 1 "from 3 to 5").
Behavioral: PCL-5 with LEC-5 questionnaire — This questionnaire will be completed during an interview with a psychologist trained in the protocol, 3 months after the sudden death.
  The PCL-5 is a 20-item self-report questionnaire that assesses the 20 symptoms of PTSD according to the DSM-V. It is associated with the LEC-5 questionnaire.
  The self-reported scale uses ratings of "0 to 4" to assess each of the symptoms.
  A threshold of 38 on the PCL-5 seems reasonable to suggest the presence of PTSD.

SUMMARY:
This study will evaluate and describe the occurrence of Acute traumatic stress and persistence of Post Traumatic Stress Disorder (PTSD) after resuscitated sudden cardiac death (SCD) in patient and relatives present during the event. The population will be composed of 40 patients: 20 with resuscitated SCD and 20 relatives. Two interviews will be performed by a psychologist within one week after resuscitated SCD and at month 3. Questionnaire Stanford Acute Stress Reaction Questionnaire (SASRQ), Life Events Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (LEC-5) and Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) will be filled during these interviews.

DETAILED DESCRIPTION:
In spite of therapeutic advances, sudden cardiac death (SCD) remains a frequent (60000/year in France) and often fatal disease (5% survival). Because it is by definition unexpected, the psychological impact on resuscitated patients and on relatives may be important. However little studies have evaluated it. Patients who later develop PTSD, generally have acute stress disorder. In patients with resuscitated sudden cardiac death, acute psychological distress is frequent and PTSD was identified in 40% of patients. Concerning relatives, Haywood (2018) call them the "forgotten patients" to emphasize the absence of recognition of his psychological trauma. PTSD was more frequent in people who were witness of the SCD vs those who were not there. Hofland et al (2018) showed that people present during resuscitation maneuvers had more acute stress than others.

This study will evaluate acute stress disorder with SASRQ scale in patients with resuscitated SCD and their relative just after the event. At 3 months, presence of PTSD will be evaluated with PCL-5 and LEC-5 in patients and their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resuscitated sudden cardiac death and/or their relative
* Patients who are fluent in French
* Patients who have given their 'no objection to participation to the research'
* Patients of both gender over 18 years
* Women with childbearing potential and effective contraception

Exclusion Criteria:

* People who are not able to give their 'no objection to participate to the research'
* People with major cognitive disorders post sudden cardiac death
* People with known psychiatric disorder
* Women who are known to be pregnant or lactating
* Person deprived of liberty by judicial or administrative decision
* People under legal protection (under the protection of a conservator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients and relatives with PTSD at months 3 post resuscitated SCD | Month 3
  The percentage of patients and relatives is determined using the PCL-5 and LEC-5 questionnaire

SECONDARY OUTCOMES:
Proportion of patients and/or relatives with acute stress disorder | Day 0
  The percentage of patients and relatives is determined using the SASRQ questionnaire
Proportion of patients and/or relatives with trauma vulnerability | Month3
  The percentage of patients and/or relatives is determined using the LEC-5 included in the PCL-5 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Banos, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France